CLINICAL TRIAL: NCT04344262
Title: Respiratory Benefits of Small Doses Muscle Relaxant in General Anesthesia
Brief Title: Small Doses Muscle Relaxant in General Anesthesia
Acronym: relaxant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Lecturer of anesthesia and surgical intensive care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: respiratory effect
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Muscle Relaxant
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated via sealed opaque envelopes into 2 groups of 30 patients each; control (C) group and minimal dose (M) group
Who Masked: Participant, Investigator
Masking Description: Basal US assessment and its repetition in the recovery room, will be done by an anesthetist who is not involved in randomization or anesthetic technique except, after ending the surgery and after dressing, he will be responsible for reversal agent injection and the extubation with recording the extubation time
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (C) group (Active Comparator): Intubating dose of muscle relaxant will be atracurium 0.5 mg/kg
  Maintenance doses of muscle relaxant will be given throughout the intraoperative period
  to maintain the Train-of-four values continuously less than 2
  Interventions: Drug: Atracurium Besylate regular dose
- minimal dose (M) group (Experimental): Intubating dose of muscle relaxant will be 0.2 mg/kg will be injected
  boluses of muscle relaxant will be given only upon complain of the surgeon and after a bolus dose of propofol 0.5 mg/kg. When required, 20% of the initial dose of muscle relaxant will be provided as a bolus to achieve this goal.
  Interventions: Drug: Atracurium Besylate minial dose

INTERVENTIONS:
Drug: Atracurium Besylate regular dose — Intubating dose of muscle relaxant will be atracurium 0.5 mg/kg
  Maintenance doses of muscle relaxant will be given throughout the intraoperative period
  to maintain the Train-of-four values continuously less than 2
  Arms: control (C) group
Drug: Atracurium Besylate minial dose — atracurium boluses of muscle relaxant given only upon complain of the surgeon and after a bolus dose of propofol 0.5 mg/kg. When required, 20% of the initial dose of muscle relaxant will be provided as a bolus to achieve this goal
  Arms: minimal dose (M) group

SUMMARY:
This study will be held to assess the effect of minimal dose muscle relaxant on postoperative pulmonary function. The time to extubation in minutes will be the primary outcome as a clinical indicator of the return of muscle power. The extubation time will be defined as the time from injecting the muscle relaxant reversing agent given when regain the train of four (TOF) ratio to 0.9 till removal of endotracheal tube.

Intraoperative surgical conditions will be assessed in the form of surgeon satisfaction and the need for more muscle relaxant boluses. Postoperative complications as desaturation (peripheral oxygen saturation (Spo2) less than 90%), the need for re-intubation or ventilation support will be recorded. Patient lung will be assessed using ultrasound-based lung aeration score. Also, the diaphragmatic and intercostal muscle function will be assessed in the early postoperative period. Immediate postoperative pulmonary function tests will be evaluated using simple spirometer. Patients will be followed up for 28 days for detection of pulmonary complications.

DETAILED DESCRIPTION:
After arrival to the operating theater, a thoracic US examination will be done using LUS dynamic re-aeration score. Patients will be randomly allocated via sealed opaque envelopes into 2 groups of 30 patients each; control (C) group and minimal dose (Min) group.

For general anesthesia; intubating dose of muscle relaxant will be injected according to the study group; in C group; atracurium 0.5 mg/kg while in min group 0.2 mg/kg will be injected. The trial for intubation will be assessed and recorded. Train-of-four (TOF) stimulation will be maintained less than 2 throughout the intraoperative period in the control group. While, in the min group, boluses of muscle relaxant will be given only upon complain of the surgeon and after a bolus dose of propofol 0.5 mg/kg. When required, 20% of the initial dose of muscle relaxant will be provided as a bolus to achieve this goal.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* aged from 20 to 50 years old
* scheduled for non-cardiothoracic surgery
* under general anesthesia
* in supine position
* after informed consent

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) score more than 3
* suspected full stomach or who will undergo intervention expected to necessitate profound muscle relaxation or dressing interferes with ultrasound (US) probe positioning
* Lung parenchymatous disease
* renal disease
* hepatic disease
* neuromuscular disease
* electrolytes imbalanc
* on medication interfere with muscle contraction
* with known allergy to any drug used in the study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-22 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The time to extubation in minutes | after injecting the muscle relaxant till removal of the tracheal tube
  the time from injecting the muscle relaxant reversing agent given when regain the train of four (TOF) ratio to 0.9 till removal of endotracheal tube

SECONDARY OUTCOMES:
Time to the first intraoperative need of muscle relaxant bolus (Atracurium), in the M group | Given intraoperatively only upon complain of the surgeon and after a bolus dose of propofol 0.5 mg/kg
  blouse of muscle relaxant given only upon complain of the surgeon and after a bolus dose of propofol 0.5 mg/kg
Total doses of propofol used in M group post-induction | intraoperatively
  a bolus dose of propofol 0.5 mg/kg given in the M group, upon complain of the surgeon and before boluses of muscle relaxant
first Postoperative day complications | after removal of the tracheal tube and for 24 hours postoperative
  desaturation (Spo2 less than 90%), need for re-intubation, need of ventilation support
lung aeration via Lung ultrasound dynamic re-aeration score | basal immmediate preoperative & with first 30 minutes postoperative
  0= normal aeration (horizontal A-lines or ≤ 2 B-lines); 1 = moderate loss of aeration (multiple B-lines, either regularly spaced (7 mm apart), or irregularly spaced and even coalescent but only visible in a limited area of the intercostal space); 2 = loss of aeration (multiple coalescent B-lines, in prevalent areas of the intercostal spaces and observed in one or several intercostal spaces); 3 = complete loss of aeration (lung consolidation, with or without air bronchograms)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Ahmed Abozeid, MD, Study Director — Faculty of Medicine - Mansoura University
Locations (1):
- Mansoura University-Emergency hospital-ICU, Al Mansurah, Egypt